CLINICAL TRIAL: NCT02713685
Title: Comparison of Combined Sciatic(Winnie's) Femoral Nerve Block, and Subarachnoid Block Anesthesia for Lower Limb Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College, Haldwani (Other)
Responsible Party: Principal Investigator, Dr Subhro Mitra, Assistant Professor, Government Medical College, Haldwani
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 294/GMC/IEC/2016
Record Dates: First submitted 2016-03-11; First posted 2016-03-21 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Anesthesia Local
Keywords: regional anesthesia; lower limb surgery; Bupivacaine
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subarachnoid block (Experimental): Subarachnoid block will be given in lateral position
  Interventions: Procedure: Subarachnoid block
- Peripheral nerve block (Active Comparator): Combined Femoral and Sciatic nerve block will be given using nerve stimulation technique
  Interventions: Procedure: combined Femoral and Sciatic nerve block

INTERVENTIONS:
Procedure: Subarachnoid block — Subarachnoid block will be given using 2.5 ml of 0.5%Bupivacaine for lower limb anesthesia
  Arms: Subarachnoid block
Procedure: combined Femoral and Sciatic nerve block — Femoral and Sciatic nerve blocks will be given using total 40 ml of 0.25%of Bupivacaine to anesthetise for lower limb surgery
  Arms: Peripheral nerve block

SUMMARY:
60 ASA grades- I, II or III patients, undergoing lower limb surgeries, will be randomly allocated in 2 groups of 30 patients each. In group S- subarachnoid block with 0.5% Bupivacaine (hyperbaric) 2.5ml will be given in lateral position and group B received femoral 3 in 1 block in supine position(with landmark technique) with 20 ml of 0.25% of Bupivacaine, followed by Sciatic block in lateral position with 20 ml of 0.25% Bupivacaine. Onset and duration of sensory and motor block, time of first analgesic requirement, VAS Scores at end of block and surgery, hemodynamic effects, patients' and surgeon's satisfaction will be evaluated.

DETAILED DESCRIPTION:
After taking approval from institutional ethics committee, 60 ASA grade - I, II, III patients will be enrolled in the study undergoing lower limb surgeries. Patients will be randomly allocated in 2 groups of 30 patients each - Group S (spinal group) and Group B (nerve block group). Informed consent shall be taken prior to procedure. Patients will also be told about VAS score for pain- 0= no pain and 10= worst imaginable pain.

In the operating room, after securing 18G IV cannula, all standard monitors will be attached (NIBP, SPO2, ECG, Temperature probe, foley's catheterization). Patients will be premedicated with inj. Ondansetron-4mg IV stat and inj. Midazolam- 1mg IV stat in both the groups before starting the procedure. Group S (SAB)- patients will be preloaded with 10mg/kg Ringer lactate. Subarachnoid block in L3-L4, L4-L5 space with 0.5% Bupivacaine (Hyperbaric)-2.5ml will be given in lateral position with involved limb in dependent position. Patient kept in same position for 15 minutes and then turned supine. Group B (peripheral nerve block)- femoral 3 in 1 block in supine position(with landmark technique) will be given with 20 ml of 0.25% of Bupivacaine followed by sciatic block in Labat's approach in lateral position with 20 ml of 0.25% Bupivacaine .

Sensory block will be evaluated using the pinprick test using 22-gauge hypodermic needle, and it will be judged adequate if there will be a complete loss of pinprick sensation at T12 in the spinal group, or in the femoral and sciatic nerve distribution in the sciatic-femoral group. Onset of Motor blockade will be taken when Bromage score 4 would have been achieved. Bromage score 1- free movement of legs and feet; 2- just able to flex knees; 3- unable to flex knees but free movement of feet; 4- unable to move legs or feet. VAS score would be assessed after the procedure and surgery. Patients' vitals will be recorded before procedure, just after the procedure and intraoperative at 5, 15 and 30 min of surgery. After completion of surgery, hemodynamic parameters would be recorded and patient would be asked about VAS score. After surgery, patient's and surgeon's satisfaction would also be evaluated as 'Yes' or 'No'. Duration of analgesia will be calculated from onset of sensory blockade to 1st requirement of analgesic (VAS score >5). Injection Diclofenac- 75mg iv infusion will be given for treatment of pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade 1/2 patients posted for unilateral lower limb orthopedic surgery

Exclusion Criteria:

* ASA grade 3/4, psychiatric patients, allergy to local anesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
duration of analgesia | 24 hours
  after surgery upto patient demands analgesia

SECONDARY OUTCOMES:
VAS score after surgery | 4 hours
  subjective VAS score after completion of surgery
onset of sensory block | 30 minutes
  sensory block will be assessed by subjective pin prick test up to achieving loss of sensation in every dermatome involved in surgery
onset of motor block | 30 minutes
  after giving block up to achievement of modified Bromage score of 4

OTHER OUTCOMES:
duration of sensory block | 4 hrs
  after block upto 2 segments regression from highest level of block
duration of motor block | 4 hrs
  after block up to start of movement of the limb
surgeon satisfaction | 4 hrs
  subjective yes/ no response
Patient satisfaction | 4 hrs
  subjective yes/no response

CONTACTS AND LOCATIONS:
Overall Officials: SUBHRO MITRA, MD, Principal Investigator — Assistant Professor
Locations (1):
- Government Medical College, Haldwani, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: Undecided